CLINICAL TRIAL: NCT04865250
Title: Exploratory Study Evaluating the Potential of Immune Signature Profiling for Predicting Response in Patients With Resectable Stage II, IIIA and Select IIIB (T3N2 Only) Non-squamous Non-Small Cell Lung Cancer (NSCLC) to Neoadjuvant ATEZOLIZUMAB Plus Carboplatin/Nab Paclitaxel
Brief Title: Predicting Response to Neoadjuvant ATEZOLIZUMAB Plus Carboplatin/Nab Paclitaxel in Resectable Non-squamous NSCLC
Acronym: iReP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Dietmar Hopp Stiftung (Other)
Responsible Party: Principal Investigator, Dirk Jäger, Professor Dr. med., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iReP
Record Dates: First submitted 2021-03-08; First posted 2021-04-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: NSCLC Stage II; NSCLC, Stage IIIA; NSCLC Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Exploratory, open-label, non-randomized, single treatment, phase II study
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): ATEZOLIZUMAB; Carboplatin; Nab-Paclitaxel
  Interventions: Drug: Atezolizumab 1200 mg abs day 1 q22 (iv)

INTERVENTIONS:
Drug: Atezolizumab 1200 mg abs day 1 q22 (iv) — Immune checkpoint blockade antibody ATEZOLIZUMAB directed against PD-L1 (Programmed death-ligand 1); Carboplatin; Nab-Paclitaxel (iv)
  Other Names: Carboplatin AUC5 day 1 q22 (iv); Nab-Paclitaxel 100 mg/m2 day 1,8,15 q22

SUMMARY:
Exploratory study evaluating the potential of immune signature profiling for predicting response in patients with resectable Stage II, IIIA and select IIIB (T3N2 only) non-squamous Non-Small Cell Lung Cancer (NSCLC) to neoadjuvant ATEZOLIZUMAB plus Carboplatin/nab Paclitaxel

Atezolizumab is given as intravenous infusion at a fixed dose of 1200 mg, day 1 of each 21-day cycle (every 3 weeks) for 3 cycles during the neoadjuvant treatment phase, Carboplatin at an initial dose of AUC (area under curve) 5 mg/mL/min, intravenously day 1 of each 21-day cycle for 3 cycles during the neoadjuvant treatment Phase, and Nab-Paclitaxel (Abraxane) at 100 mg/m2, intravenously day 1, 8 and 15 of each 21-day cycle for 3 cycles during the neoadjuvant treatment phase. Surgery after the 3rd cycle Atezolizumab / Carboplatin / Nab-Paclitaxel is standard procedure.

DETAILED DESCRIPTION:
In early stages of non-small cell lung cancer (NSCLC), surgical treatment with curative intent is the treatment of choice. Adjuvant chemotherapy is standard of care for fully resected stage II, IIIA, or select IIIB [T3N2] NSCLC to improve survival outcome as compared to surgery alone. Neoadjuvant platinum-based chemotherapy has become a widely accepted alternative therapy. Chemotherapy regimens used in the adjuvant and neoadjuvant settings consist of platinum-based doublets. With the successful development of cancer immunotherapy in advanced NSCLC, several (neo)adjuvant studies of anti-PD-1/PD-L1 inhibitors are currently being conducted in resectable early-stage NSCLC.

The IREP study explores neoadjuvant immunochemotherapy with three cycles of atezolizumab, carboplatin and nab-paclitaxel in patients with histologically confirmed and resectable non-squamous NSCLC Stage II, IIIA or select IIIB (T3N2 only). The primary endpoint of the study is the Major Pathologic Response (MPR) rate (≤10% residual viable tumor cells) at surgery. Secondary endpoints include EFS and OS, safety endpoints as well as analyses of molecular and immunological biomarkers that are predictive of response to the neoadjuvant immunochemotherapy treatment.

Atezolizumab is given as intravenous infusion at a fixed dose of 1200 mg day 1, carboplatin at an initial dose of AUC 5 mg/mL/min intravenously day 1 and nab-paclitaxel at 100 mg/m2 intravenously day 1, 8 and 15 of each 21-day cycle (every 3 weeks) for 3 cycles during the neoadjuvant treatment phase. Subsequent surgery is standard procedure with standard lobectomy / bi-lobectomy with systematic lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, patients age ≥ 18-year-old including, signed and dated
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Histologically confirmed NSCLC of non-squamous histology, cStage II, IIIA or select IIIB (T3N2 only); for T-status ≤ T3 allowed; for N2 patients only IIIa1-3 Robinson classification allowed
* Deemed surgically resectable with curative intent by an attending thoracic surgeon after adequate staging including PET-CT (positron emission tomography)
* Adequate lung and cardiac function for intended lung resection according to German S3 regulation
* Radiologically measurable disease as defined by response evaluation criteria in solid tumors RECIST v1.1
* Sufficient availability of the tissue sample from primary tumor before start of neoadjuvant treatment
* Females of child-bearing potential must agree to use, and be able to comply with, effective contraception (</=1% failure rate annually) without interruption, 28 days prior to starting therapy (including dose interruptions), and while on study medication or for a period of 120 days after the last dose of study medication
* Females must have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy.
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following treatment discontinuation, even if he has undergone a successful vasectomy.
* adequate renal, hepatic, and bone marrow function as defined below

  * Absolute neutrophil count (ANC) > 1500/μl
  * Platelet count ≥ 100000/μl
  * Hemoglobin ≥ 9 g/dl (can be post-transfusion)
  * International normalized ratio (INR) ≤ 1.4 in patients not receiving anticoagulation; for patients receiving respective anticoagulation an INR ≤3.0 allowed
  * Activated partial thromboplastin time (aPTT) ≤ 1.5 times upper limit of normal (ULN) in patients not receiving anticoagulation; for patients receiving respective anticoagulation a PTT ≤2.5 ULN allowed
  * Bilirubin < 1.5 times ULN (for patients with known Gilbert disease Bilirubin ≤ 3 times ULN allowed)
  * ALT and AST < 2.5 times ULN
  * Creatinine ≤ 1.5 ULN or calculated creatinine clearance > 60 ml/min for subjects with creatinine levels > 1.5 ULN; for patients meeting the criterion of creatinine ≤ 1.5 ULN also a calculated creatinine clearance of > 30 ml/min is mandatory

Exclusion Criteria:

* Illness or condition that may interfere with a patient's capacity to understand, follow, and/or comply with study procedures
* Treatment in any other clinical trial within 30 days before screening.
* NSCLC Stage cT4
* NSCLC stage cN3 or cN2 IIIA4 (bulky or fixed multi-station N2 disease) according to Robinson classification
* NSCLC of squamous cell histology
* Any prior therapy for lung cancer (including systemic therapy, radiotherapy or major surgery)
* Malignancies other than NSCLC within 5 years prior to study inclusion with the exception of malignancies with a negligible risk of metastasis or death (5-year OS > 90%) like localized prostate cancer, ductal carcinoma in situ, adequately treated carcinoma in situ of the cervix, Stage I uterine cancer or non-melanoma skin carcinoma
* History of allogeneic tissue / solid organ transplant or allogeneic stem cell transplantation
* Patients with active hepatitis B or C infections or a history of HIV infection
* Pregnant or lactating women
* Active autoimmune disease or history of severe autoimmune disease or immunodeficiency or a syndrome that requires systemic steroids or immunosuppressive agents
* The following exceptions are granted:

  * patients with vitiligo, eczema, lichen simplex or resolved childhood asthma/atopy
  * subjects requiring intermittent use of bronchodilatators or local steroid injections
  * patients with hypothyroidism stable on hormone replacement
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, and anti-tumor necrosis factor (anti-TNF) agents) within 2 weeks prior to Cycle 1, Day 1 (except low-dose steroids for adrenal failure or emesis prophylaxis)
* History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia, drug-induced pneumonitis, or evidence of active pneumonitis on screening chest Computed Tomography (CT) scan
* Prior treatment with cluster of differentiation 137 (CD137) agonist or immune checkpoint blockade therapies, anti-programmed-death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibody
* Live vaccine within 30 days prior to first dose of trial treatment
* Cerebrovascular accident within the past 6 months
* Severe infection or significant traumatic injury within the past 4 weeks
* Clinically significant history of cardiovascular disease, including any of the following:

  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class II, III-IV congestive heart failure
  * Poorly controlled cardiac arrhythmia despite medication, except rate-controlled atrial fibrillation
* Known allergy or hypersensitivity to any component of the chemotherapy regimen Patients who have been incarcerated or involuntarily institutionalized by court order or by the authorities, as well as patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Response to neoadjuvant immunochemotherapy with ATEZOLIZUMAB, Carboplatin and nab-Paclitaxel | up to 5 months (after 9 weeks of neoadjuvant immunochemotherapy (3 cycles with 21 days per cycle) + surgery (4-8 additional weeks after completion of neoadjuvant immunochemotherapy)
  determined by Major Pathologic Response (MPR) (≤10% residual viable tumor cells) (pathologic regression grading according to Junker criteria) rate

SECONDARY OUTCOMES:
Response rate according to RECIST 1.1 criteria | pre-surgery after completion of neoadjuvant immunochemotherapy
  determined by Δ tumor size and Δ lymph node size
Response rate as determined by Δ PETactivity | pre-surgery after completion of neoadjuvant immunochemotherapy
  determined by standardized uptake value [SUV] (standard uptake value)
Event-free survival (EFS) | up to 29 months after study inclusion; calculated from start of 1st cycle of neoadjuvant treatment, thus including three 21 day cycles+surgery, follow-up for 24 months after end of treatment visit; end of treatment visit takes place 6 weeks after surgery
  time to any of the following events, whichever occurs first: progression of disease prior to surgery as defined by RECIST v1.1, local or distant disease recurrence, or death due to any cause
Overall survival (OS) | up to 29 months after study inclusion; calculated from start of 1st cycle of neoadjuvant treatment, thus including three 21 day cycles+surgery, follow-up for 24 months after end of treatment visit; end of treatment visit takes place 6 weeks after surgery
  time to death due to any cause
Number of patients attaining surgery as planned | up to 5 months
  number of patients attaining surgery divided by the total number of patients included

CONTACTS AND LOCATIONS:
Locations (1):
- Thoraxklinik Heidelberg gGmbH, Heidelberg, BaWü, Germany

IPD SHARING:
Plan to Share IPD: No